CLINICAL TRIAL: NCT04168645
Title: Inpatient Cognitive-Behavioral Therapy to Reduce Suicide Risk Post-Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, David Tolin, Director, Anxiety Disorders Center, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHC-2019-0163
Record Dates: First submitted 2019-11-09; First posted 2019-11-19 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Suicide, Attempted
MeSH Terms: conditions — Suicide, Attempted | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned (using a computer-generated randomization schedule) to either BCBT or TAU using stratified block randomization on Substance Use Disorder (SUD). We expect, based on pilot data analyses, that approximately two-thirds of patients in each group will be diagnosed with SUD.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Presence of SUD with BCBT (Experimental): Patients diagnosed with SUD who are randomly assigned to receive BCBT will participate in all aspects of their prescribed treatment plan (i.e., TAU) and will receive up to 4 sessions of CBT (depending on length of stay), lasting 1.5 hours for the first session and 1 hour for the remaining sessions.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Presence of SUD with TAU (No Intervention): Patients diagnosed with SUD who are randomly assigned to receive TAU will participate in all aspects of the prescribed treatment plan given by the inpatient unit.
- Absence of SUD with BCBT (Experimental): Patients without SUD who are randomly assigned to receive BCBT will participate in all aspects of their prescribed treatment plan (i.e., TAU) and will receive up to 4 sessions of BCBT (depending on length of stay), lasting 1.5 hours for the first session and 1 hour for the remaining sessions.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Absence of SUD with TAU (No Intervention): Patients without SUD who are randomly assigned to receive TAU will participate in all aspects of the prescribed treatment plan given by the inpatient unit.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Up to 4 sessions of BCBT (depending on length of stay) will be provided. The first session lasts 1.5 hours and subsequent sessions are 1 hour.
  Arms: Absence of SUD with BCBT; Presence of SUD with BCBT

SUMMARY:
The goal of this randomized-controlled trial is to determine whether adding brief cognitive-behavioral therapy for suicide prevention (BCBT) to inpatient treatment improves suicide-related outcomes after the person leaves the hospital. The study will also determine whether being diagnosed with a substance use disorder impacts these outcomes. Participants will either receive treatment as usual or treatment as usual plus up to four sessions of BCBT during their inpatient stay. They will complete monthly follow-up assessments for six months after leaving the hospital.

DETAILED DESCRIPTION:
Although inpatient treatment provides immediate stabilization and crisis management for suicidal patients, the risk of suicide post-discharge is substantial, with approximately one third of all suicides by individuals with mental disorders occurring in the 90 days following hospitalization. These data highlight the importance of establishing an empirically-supported inpatient treatment for suicide prevention. Cognitive behavioral therapy (CBT) is a strong candidate, given that CBT reduces risk in suicidal outpatients. In addition, an open trial was completed that 1) adapted the strongest outpatient CBT protocol for an inpatient setting, 2) demonstrated high levels of feasibility and acceptability, and 3) obtained preliminary estimates of efficacy. The objective here is to conduct a largescale randomized controlled trial (RCT) comparing brief cognitive-behavioral therapy for suicide prevention (BCBT) (n = 100) to treatment as usual (TAU, n = 100) to firmly establish efficacy and collect pilot data on treatment implementation metrics. This study aims to determine the efficacy of inpatient BCBT on suicidal behavior, suicidal ideation/intent, and readmission post-treatment and over a 6-month follow-up period. The central hypothesis, based on strong outpatient data, is that inpatient BCBT will reduce suicidal behavior, suicidal ideation/intent, and inpatient readmission over 6 months post-discharge, compared to TAU. Participants will be recruited after inpatient admission following a suicide attempt or with suicidal ideation and plan with suicide attempt within the previous two years. Participants assigned to the BCBT condition will receive four BCBT sessions in addition to treatment as usual. Assessments will occur at intake, discharge, and monthly for six months post-discharge. The proposed study will inform best practices treatment for hospitalized suicidal patients by establishing for the first time, and ultimately disseminating, an empirically-validated inpatient treatment for suicide prevention.

ELIGIBILITY:
Inclusion Criteria:

* Any Gender
* Age 18-65 inclusive
* Fluent in English (speaking, reading, and writing)
* Having made a suicide attempt within one week preceding admission or suicidal ideation and plan on admissions along with suicide attempt within previous two years. Admission will be defined as admission to either the medical floor (in cases where medical stabilization is required prior to transfer to psychiatric inpatient facility) or to psychiatric inpatient facility (in cases where medical stabilization is not required). A suicide attempt will be defined as behavior that is self-directed and deliberately results in injury or the potential for injury to oneself for which there is evidence, whether explicit or implicit, of intent to die.

Exclusion Criteria:

* Age <18 or ≥66 years old
* History of schizophrenia or schizoaffective disorder
* History of intellectual disability or organic brain illness
* Active mania or other psychiatric or medical condition that would preclude informed consent or participation in the trial, in the investigator's opinion
* ECT included on patient's inpatient treatment plan. Patients who are referred for ECT after starting the study will be withdrawn from the study.
* Discharge expected within four business days of attending approval.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F Tolin, Ph.D., Principal Investigator — Institute of Living/Hartford Hospital
Locations (1):
- Institute of Living/Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diefenbach GJ, Lord KA, Stubbing J, Rudd MD, Levy HC, Worden B, Sain KS, Bimstein JG, Rice TB, Everhardt K, Gueorguieva R, Tolin DF. Brief Cognitive Behavioral Therapy for Suicidal Inpatients: A Randomized Clinical Trial. JAMA Psychiatry. 2024 Dec 1;81(12):1177-1186. doi: 10.1001/jamapsychiatry.2024.2349. PMID 39259550
- [Derived] Stubbing J, Tolin DF, Sain KS, Everhardt K, Rudd MD, Diefenbach GJ. Borderline Personality Traits Do Not Moderate the Relationship Between Depression, Beliefs, and Suicidal Thoughts and Behaviors. Arch Suicide Res. 2025 Jan-Mar;29(1):223-237. doi: 10.1080/13811118.2024.2345168. Epub 2024 Apr 29. PMID 38683542
- [Derived] Diefenbach GJ, Stubbing J, Rice TB, Lord KA, Rudd MD, Tolin DF. Uncovering the role of substance use in suicide attempts using a mixed-methods approach. Suicide Life Threat Behav. 2024 Feb;54(1):70-82. doi: 10.1111/sltb.13019. Epub 2023 Nov 21. PMID 37987548
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Presence of SUD With BCBT | Presence of SUD With TAU | Absence of SUD With BCBT | Absence of SUD With TAU
Started | 62 | 65 | 41 | 45
Intent to Treat | 56 | 64 | 38 | 42
Completed | 30 | 33 | 23 | 28
Not Completed | 32 | 32 | 18 | 17
Not completed — Lost to Follow-up | 23 | 28 | 15 | 12
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 2 | 2 | 2
Not completed — Administrative Withdrawal | 3 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Presence of SUD With BCBT | Presence of SUD With TAU | Absence of SUD With BCBT | Absence of SUD With TAU | Total
Number analyzed (Participants) | 62 | 65 | 41 | 45 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.00 (11.70) | 32.68 (11.71) | 33.22 (14.28) | 32.09 (14.01) | 33.04 (12.67)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: There was missing gender identity data for two participants.
  Participants
    Gender Identity: Male | 24 | 32 | 13 | 12 | 81
    Gender Identity: Female | 30 | 28 | 23 | 26 | 107
    Gender Identity: Trans Male | 3 | 1 | 0 | 1 | 5
    Gender Identity: Trans Female | 2 | 1 | 1 | 2 | 6
    Gender Identity: Genderqueer/Gender Non-Conforming | 2 | 3 | 2 | 4 | 11
    Gender Identity: Do Not Identify As Any of These Options | 0 | 0 | 0 | 0 | 0
    Gender Identity: Prefer Not to Answer | 1 | 0 | 0 | 0 | 1
    Gender Identity: Missing | 0 | 0 | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth. Population: There was missing sex assigned at birth data for one participant.
  Participants
    number analyzed (Participants) | 61 | 65 | 41 | 45 | 212
    Female | 34 | 31 | 27 | 30 | 122
    Male | 27 | 34 | 14 | 15 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 19 | 6 | 10 | 51
  Not Hispanic or Latino | 45 | 43 | 30 | 35 | 153
  Unknown or Not Reported | 1 | 3 | 5 | 0 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 42 | 37 | 26 | 28 | 133
  Race: Black or African American | 6 | 9 | 7 | 8 | 30
  Race: Asian | 0 | 0 | 1 | 1 | 2
  Race: Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 1 | 1
  Race: American Indian or Alaskan Native | 1 | 1 | 1 | 0 | 3
  Race: Multiracial | 4 | 5 | 0 | 0 | 9
  Race: Other | 7 | 12 | 4 | 6 | 29
  Race: Prefer Not to Answer | 2 | 1 | 2 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 65 | 41 | 45 | 213
Columbia Suicide Severity Rating Scale Lifetime Actual Suicide Attempts [Median (Standard Deviation); unit: Number of Attempts] | 2 (9.21) | 3 (3.71) | 2 (2.44) | 2 (2.43) | 2 (5.67)
Columbia Suicide Severity Rating Scale Lifetime Interrupted Suicide Attempts [Median (Standard Deviation); unit: Number of Attempts] | 0.00 (1.93) | 0.00 (1.97) | 0.00 (0.62) | 0.00 (0.50) | 0.00 (1.55)
Columbia Suicide Severity Rating Scale Lifetime Aborted Suicide Attempts [Median (Standard Deviation); unit: Number of Attempts] | 0.00 (4.11) | 0.00 (6.86) | 0.00 (3.82) | 0.00 (30.46) | 0.00 (14.80)
Columbia Suicide Severity Rating Scale Lifetime Preparatory Events [Median (Standard Deviation); unit: Number of Preparatory Events] | 0.00 (7.99) | 0.00 (25.55) | 0.00 (11.71) | 1.00 (72.72) | 0.00 (37.31)
Columbia Suicide Severity Rating Scale Past Month Most Severe Ideation [Count of Participants; unit: Participants] — Most severe suicidal ideation in the past month indicated by the respondent.
  Participants
    Active Suicidal Ideation with Any Methods | 0 | 2 | 0 | 1 | 3
    Active Suicidal Ideation with Some Intent to Act | 0 | 2 | 0 | 0 | 2
    Active Suicidal Ideation with Specific Plan | 62 | 61 | 41 | 44 | 208
Columbia Suicide Severity Rating Scale Past Month Suicidal Ideation Intensity [Mean (Standard Deviation); unit: units on a scale] — Scores on the Columbia Suicide Severity Rating Scale range from 0 to 25 with higher scores representing more severe suicidal ideation
  units on a scale | 19.18 (3.02) | 18.17 (3.68) | 18.05 (3.41) | 18.04 (3.06) | 18.42 (3.33)
Columbia Suicide Severity Rating Scale Lifetime Actual Suicide Attempts [Count of Participants; unit: Participants] — Number of participants endorsing lifetime actual suicide attempts on Columbia Suicide Severity Rating Scale
  Participants | 60 | 65 | 39 | 41 | 205
Columbia Suicide Severity Rating Scale Lifetime Interrupted Suicide Attempts [Count of Participants; unit: Participants] | 24 | 19 | 12 | 11 | 66
Columbia Suicide Severity Rating Scale Lifetime Aborted Suicide Attempts [Count of Participants; unit: Participants] | 16 | 20 | 12 | 18 | 66
Columbia Suicide Severity Rating Scale Lifetime Preparatory Events [Count of Participants; unit: Participants] | 24 | 32 | 13 | 23 | 92

OUTCOME MEASURES:

1. Primary Outcome: Columbia Suicide Severity Rating Scale Number of Participants Reporting Presence of Suicidal Behaviors
Description: Suicidal behavior will be assessed using the Columbia Suicide Severity Rating Scale (C-SSRS), a widely used suicide assessment measure. Several suicidal behaviors are assessed on the C-SSRS including the presence or absence of each of the following: suicide attempt, interrupted attempt, aborted attempt, and preparatory acts or behaviors. Scores reflect the number of participants with the presence of the suicide behavior.
Time Frame: Assessed at completion of inpatient treatment (average of 12 days), and on a monthly basis for 6 months follow-up.
Population: Data were missing due to attrition.
Measure: Count of Participants; unit: Participants
Arm/Group | Presence of SUD With BCBT | Presence of SUD With TAU | Absence of SUD With BCBT | Absence of SUD With TAU
Number analyzed (Participants) | 53 | 57 | 38 | 41
Participants
  Actual Suicide Attempt at Post-treatment | 1 | 1 | 0 | 0
  Actual Suicide Attempt at Follow-up 1: number analyzed (Participants) | 45 | 48 | 34 | 37
  Actual Suicide Attempt at Follow-up 1 | 1 | 4 | 0 | 2
  Actual Suicide Attempt at Follow-up 2: number analyzed (Participants) | 42 | 47 | 30 | 35
  Actual Suicide Attempt at Follow-up 2 | 3 | 4 | 0 | 3
  Actual Suicide Attempt at Follow-up 3: number analyzed (Participants) | 38 | 45 | 29 | 32
  Actual Suicide Attempt at Follow-up 3 | 1 | 4 | 0 | 2
  Actual Suicide Attempt at Follow-up 4: number analyzed (Participants) | 36 | 39 | 27 | 34
  Actual Suicide Attempt at Follow-up 4 | 0 | 2 | 0 | 3
  Actual Suicide Attempt at Follow-up 5: number analyzed (Participants) | 34 | 37 | 24 | 31
  Actual Suicide Attempt at Follow-up 5 | 2 | 3 | 2 | 1
  Actual Suicide Attempt at Follow-up 6: number analyzed (Participants) | 30 | 33 | 23 | 28
  Actual Suicide Attempt at Follow-up 6 | 1 | 2 | 0 | 0
  Interrupted Suicide Attempt at Post-treatment | 0 | 0 | 0 | 1
  Interrupted Suicide Attempt at Follow-up 1: number analyzed (Participants) | 45 | 48 | 34 | 37
  Interrupted Suicide Attempt at Follow-up 1 | 0 | 2 | 0 | 0
  Interrupted Suicide Attempt at Follow-up 2: number analyzed (Participants) | 42 | 47 | 30 | 35
  Interrupted Suicide Attempt at Follow-up 2 | 0 | 2 | 0 | 0
  Interrupted Suicide Attempt at Follow-up 3: number analyzed (Participants) | 38 | 45 | 29 | 32
  Interrupted Suicide Attempt at Follow-up 3 | 2 | 1 | 0 | 1
  Interrupted Suicide Attempt at Follow-up 4: number analyzed (Participants) | 36 | 39 | 27 | 34
  Interrupted Suicide Attempt at Follow-up 4 | 0 | 1 | 0 | 0
  Interrupted Suicide Attempt at Follow-up 5: number analyzed (Participants) | 34 | 37 | 24 | 31
  Interrupted Suicide Attempt at Follow-up 5 | 0 | 1 | 0 | 0
  Interrupted Suicide Attempt at Follow-up 6: number analyzed (Participants) | 30 | 33 | 23 | 28
  Interrupted Suicide Attempt at Follow-up 6 | 0 | 1 | 0 | 0
  Aborted Suicide Attempt at Post-treatment | 1 | 1 | 0 | 2
  Aborted Suicide Attempt at Follow-up 1: number analyzed (Participants) | 46 | 48 | 34 | 37
  Aborted Suicide Attempt at Follow-up 1 | 1 | 1 | 0 | 0
  Aborted Suicide Attempt at Follow-up 2: number analyzed (Participants) | 42 | 47 | 30 | 35
  Aborted Suicide Attempt at Follow-up 2 | 1 | 1 | 0 | 0
  Aborted Suicide Attempt at Follow-up 3: number analyzed (Participants) | 38 | 45 | 29 | 32
  Aborted Suicide Attempt at Follow-up 3 | 0 | 2 | 0 | 1
  Aborted Suicide Attempt at Follow-up 4: number analyzed (Participants) | 36 | 39 | 27 | 34
  Aborted Suicide Attempt at Follow-up 4 | 0 | 0 | 0 | 2
  Aborted Suicide Attempt at Follow-up 5: number analyzed (Participants) | 34 | 37 | 24 | 31
  Aborted Suicide Attempt at Follow-up 5 | 1 | 0 | 0 | 0
  Aborted Suicide Attempt at Follow-up 6: number analyzed (Participants) | 29 | 33 | 23 | 28
  Aborted Suicide Attempt at Follow-up 6 | 1 | 0 | 2 | 0
  Preparatory Events at Post-treatment: number analyzed (Participants) | 53 | 57 | 37 | 41
  Preparatory Events at Post-treatment | 1 | 1 | 1 | 2
  Preparatory Events at Follow-up 1: number analyzed (Participants) | 46 | 48 | 34 | 37
  Preparatory Events at Follow-up 1 | 1 | 3 | 0 | 4
  Preparatory Events at Follow-up 2: number analyzed (Participants) | 42 | 47 | 30 | 35
  Preparatory Events at Follow-up 2 | 0 | 1 | 1 | 2
  Preparatory Events at Follow-up 3: number analyzed (Participants) | 38 | 45 | 29 | 32
  Preparatory Events at Follow-up 3 | 0 | 1 | 2 | 2
  Preparatory Events at Follow-up 4: number analyzed (Participants) | 36 | 39 | 27 | 34
  Preparatory Events at Follow-up 4 | 1 | 2 | 2 | 0
  Preparatory Events at Follow-up 5: number analyzed (Participants) | 34 | 37 | 24 | 31
  Preparatory Events at Follow-up 5 | 1 | 0 | 0 | 1
  Preparatory Events at Follow-up 6: number analyzed (Participants) | 30 | 33 | 23 | 28
  Preparatory Events at Follow-up 6 | 1 | 0 | 2 | 0

2. Primary Outcome: Columbia Suicide Severity Rating Scale Number of Suicidal Behaviors
Description: Suicidal behavior will be assessed using the Columbia Suicide Severity Rating Scale (C-SSRS), a widely used suicide assessment measure. Several suicidal behaviors are assessed on the C-SSRS including the presence or absence of each of the following: suicide attempt, interrupted attempt, aborted attempt, and preparatory acts or behaviors. Scores on this scale reflect the median number of each behavior.
Time Frame: Assessed at completion of inpatient treatment (average of 12 days), and on a monthly basis for 6 months follow-up.
Population: Data were missing due to attrition.
Measure: Median (Standard Deviation); unit: Number of Events
Arm/Group | Presence of SUD With BCBT | Presence of SUD With TAU | Absence of SUD With BCBT | Absence of SUD With TAU
Number analyzed (Participants) | 53 | 57 | 39 | 41
Number of Events
  Actual Suicide Attempt at Post-treatment | 0.00 (0.14) | 0.00 (0.13) | 0.00 (0.00) | 0.00 (0.00)
  Actual Suicide Attempt at Follow-up 1: number analyzed (Participants) | 45 | 48 | 34 | 37
  Actual Suicide Attempt at Follow-up 1 | 0.00 (0.15) | 0.00 (0.28) | 0.00 (0.00) | 0.00 (0.36)
  Actual Suicide Attempt at Follow-up 2: number analyzed (Participants) | 42 | 47 | 30 | 35
  Actual Suicide Attempt at Follow-up 2 | 0.00 (0.26) | 0.00 (0.80) | 0.00 (0.00) | 0.00 (0.40)
  Actual Suicide Attempt at Follow-up 3: number analyzed (Participants) | 38 | 45 | 29 | 32
  Actual Suicide Attempt at Follow-up 3 | 0.00 (0.16) | 0.00 (1.69) | 0.00 (0.00) | 0.00 (0.25)
  Actual Suicide Attempt at Follow-up 4: number analyzed (Participants) | 36 | 39 | 27 | 34
  Actual Suicide Attempt at Follow-up 4 | 0.00 (0.00) | 0.00 (0.22) | 0.00 (0.00) | 0.00 (0.29)
  Actual Suicide Attempt at Follow-up 5: number analyzed (Participants) | 34 | 37 | 24 | 31
  Actual Suicide Attempt at Follow-up 5 | 0.00 (0.38) | 0.00 (0.48) | 0.00 (0.83) | 0.00 (0.18)
  Actual Suicide Attempt at Follow-up 6: number analyzed (Participants) | 30 | 33 | 23 | 28
  Actual Suicide Attempt at Follow-up 6 | 0.00 (0.18) | 0.00 (0.38) | 0.00 (0.00) | 0.00 (0.00)
  Interrupted Suicide Attempt at Post-treatment | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.16)
  Interrupted Suicide Attempt at Follow-up 1: number analyzed (Participants) | 45 | 48 | 34 | 37
  Interrupted Suicide Attempt at Follow-up 1 | 0.00 (0.00) | 0.00 (0.32) | 0.00 (0.00) | 0.00 (0.00)
  Interrupted Suicide Attempt at Follow-up 2: number analyzed (Participants) | 42 | 47 | 30 | 35
  Interrupted Suicide Attempt at Follow-up 2 | 0.00 (0.00) | 0.00 (0.20) | 0.00 (0.00) | 0.00 (0.00)
  Interrupted Suicide Attempt at Follow-up 3: number analyzed (Participants) | 38 | 45 | 29 | 32
  Interrupted Suicide Attempt at Follow-up 3 | 0.00 (0.36) | 0.00 (0.15) | 0.00 (0.00) | 0.00 (0.18)
  Interrupted Suicide Attempt at Follow-up 4: number analyzed (Participants) | 36 | 39 | 27 | 34
  Interrupted Suicide Attempt at Follow-up 4 | 0.00 (0.00) | 0.00 (0.16) | 0.00 (0.00) | 0.00 (0.00)
  Interrupted Suicide Attempt at Follow-up 5: number analyzed (Participants) | 34 | 37 | 24 | 31
  Interrupted Suicide Attempt at Follow-up 5 | 0.00 (0.00) | 0.00 (0.16) | 0.00 (0.00) | 0.00 (0.00)
  Interrupted Suicide Attempt at Follow-up 6: number analyzed (Participants) | 30 | 33 | 23 | 28
  Interrupted Suicide Attempt at Follow-up 6 | 0.00 (0.00) | 0.00 (0.17) | 0.00 (0.00) | 0.00 (0.00)
  Aborted Suicide Attempt at Post-treatment | 0.00 (0.14) | 0.00 (0.13) | 0.00 (0.00) | 0.00 (0.35)
  Aborted Suicide Attempt at Follow-up 1: number analyzed (Participants) | 46 | 48 | 34 | 37
  Aborted Suicide Attempt at Follow-up 1 | 0.00 (0.15) | 0.00 (0.14) | 0.00 (0.00) | 0.00 (0.00)
  Aborted Suicide Attempt at Follow-up 2: number analyzed (Participants) | 42 | 47 | 30 | 35
  Aborted Suicide Attempt at Follow-up 2 | 0.00 (0.15) | 0.00 (0.15) | 0.00 (0.00) | 0.00 (0.00)
  Aborted Suicide Attempt at Follow-up 3: number analyzed (Participants) | 38 | 45 | 29 | 32
  Aborted Suicide Attempt at Follow-up 3 | 0.00 (0.00) | 0.00 (0.21) | 0.00 (0.00) | 0.00 (0.35)
  Aborted Suicide Attempt at Follow-up 4: number analyzed (Participants) | 36 | 39 | 27 | 34
  Aborted Suicide Attempt at Follow-up 4 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.24)
  Aborted Suicide Attempt at Follow-up 5: number analyzed (Participants) | 34 | 37 | 24 | 31
  Aborted Suicide Attempt at Follow-up 5 | 0.00 (0.34) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Aborted Suicide Attempt at Follow-up 6: number analyzed (Participants) | 30 | 33 | 23 | 28
  Aborted Suicide Attempt at Follow-up 6 | 0.00 (0.18) | 0.00 (0.00) | 0.00 (0.29) | 0.00 (0.00)
  Preparatory Events at Post-treatment: number analyzed (Participants) | 53 | 57 | 37 | 41
  Preparatory Events at Post-treatment | 0.00 (0.27) | 0.00 (0.13) | 0.00 (0.33) | 0.00 (0.22)
  Preparatory Events at Follow-up 1: number analyzed (Participants) | 46 | 48 | 34 | 37
  Preparatory Events at Follow-up 1 | 0.00 (0.15) | 0.00 (1.23) | 0.00 (0.00) | 0.00 (0.31)
  Preparatory Events at Follow-up 2: number analyzed (Participants) | 42 | 47 | 30 | 35
  Preparatory Events at Follow-up 2 | 0.00 (0.00) | 0.00 (0.15) | 0.00 (0.18) | 0.00 (0.37)
  Preparatory Events at Follow-up 3: number analyzed (Participants) | 38 | 45 | 29 | 32
  Preparatory Events at Follow-up 3 | 0.00 (0.00) | 0.00 (0.15) | 0.00 (0.58) | 0.00 (0.25)
  Preparatory Events at Follow-up 4: number analyzed (Participants) | 36 | 39 | 27 | 34
  Preparatory Events at Follow-up 4 | 0.00 (0.17) | 0.00 (0.22) | 0.00 (0.27) | 0.00 (0.00)
  Preparatory Events at Follow-up 5: number analyzed (Participants) | 34 | 37 | 24 | 31
  Preparatory Events at Follow-up 5 | 0.00 (0.51) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.18)
  Preparatory Events at Follow-up 6: number analyzed (Participants) | 30 | 33 | 23 | 28
  Preparatory Events at Follow-up 6 | 0.00 (0.18) | 0.00 (0.00) | 0.00 (0.29) | 0.00 (0.00)

3. Primary Outcome: The Number of Participants Reporting Columbia Suicide Severity Rating Scale Suicidal Ideation Categories as Most Severe
Description: The number of participants endorsing each category as the highest (most severe) suicidal ideation category on the Columbia Suicide Severity Rating Scale (C-SSRS) ranging from 1-5, with 5 being the most severe type of suicidal ideation.
Time Frame: Assessed at completion of inpatient treatment (average of 12 days), and on a monthly basis for 6 months follow-up.
Population: Data were missing due to attrition.
Measure: Count of Participants; unit: Participants
Arm/Group | Presence of SUD With BCBT | Presence of SUD With TAU | Absence of SUD With BCBT | Absence of SUD With TAU
Number analyzed (Participants) | 53 | 56 | 38 | 41
Participants
  Most Severe Ideation at Post-treatment: None | 31 | 21 | 20 | 15
  Most Severe Ideation at Post-treatment: Wish to be Dead | 7 | 16 | 8 | 4
  Most Severe Ideation at Post-treatment: Non-Specific Active Suicidal Thoughts | 2 | 3 | 3 | 1
  Most Severe Ideation at Post-treatment: Active Suicidal Ideation with Any Methods | 5 | 5 | 2 | 9
  Most Severe Ideation at Post-treatment: Active Suicidal Ideation with Some Intent to Act | 1 | 3 | 0 | 2
  Most Severe Ideation at Post-treatment: Active Suicidal Ideation with Specific Plan | 7 | 8 | 5 | 10
  Most Severe Ideation at Follow-up 1: number analyzed (Participants) | 46 | 47 | 34 | 36
  Most Severe Ideation at Follow-up 1: None | 32 | 23 | 16 | 12
  Most Severe Ideation at Follow-up 1: Wish to be Dead | 3 | 11 | 8 | 11
  Most Severe Ideation at Follow-up 1: Non-Specific Active Suicidal Thoughts | 0 | 1 | 6 | 5
  Most Severe Ideation at Follow-up 1: Active Suicidal Ideation with Any Methods | 4 | 4 | 1 | 3
  Most Severe Ideation at Follow-up 1: Active Suicidal Ideation with Some Intent to Act | 2 | 0 | 1 | 1
  Most Severe Ideation at Follow-up 1: Active Suicidal Ideation with Specific Plan | 5 | 8 | 2 | 4
  Most Severe Ideation at Follow-up 2: number analyzed (Participants) | 42 | 47 | 30 | 35
  Most Severe Ideation at Follow-up 2: None | 28 | 24 | 14 | 18
  Most Severe Ideation at Follow-up 2: Wish to be Dead | 4 | 10 | 9 | 8
  Most Severe Ideation at Follow-up 2: Non-Specific Active Suicidal Thoughts | 0 | 2 | 1 | 2
  Most Severe Ideation at Follow-up 2: Active Suicidal Ideation with Any Methods | 4 | 4 | 4 | 2
  Most Severe Ideation at Follow-up 2: Active Suicidal Ideation with Some Intent to Act | 1 | 1 | 0 | 0
  Most Severe Ideation at Follow-up 2: Active Suicidal Ideation with Specific Plan | 5 | 6 | 2 | 5
  Most Severe Ideation at Follow-up 3: number analyzed (Participants) | 37 | 45 | 29 | 32
  Most Severe Ideation at Follow-up 3: None | 24 | 25 | 16 | 18
  Most Severe Ideation at Follow-up 3: Wish to be Dead | 7 | 10 | 8 | 8
  Most Severe Ideation at Follow-up 3: Non-Specific Active Suicidal Thoughts | 0 | 1 | 0 | 0
  Most Severe Ideation at Follow-up 3: Active Suicidal Ideation with Any Methods | 2 | 3 | 1 | 0
  Most Severe Ideation at Follow-up 3: Active Suicidal Ideation with Some Intent to Act | 0 | 0 | 0 | 2
  Most Severe Ideation at Follow-up 3: Active Suicidal Ideation with Specific Plan | 4 | 6 | 4 | 4
  Most Severe Ideation at Follow-up 4: number analyzed (Participants) | 37 | 39 | 27 | 34
  Most Severe Ideation at Follow-up 4: None | 31 | 21 | 15 | 15
  Most Severe Ideation at Follow-up 4: Wish to be Dead | 4 | 12 | 9 | 8
  Most Severe Ideation at Follow-up 4: Non-Specific Active Suicidal Thoughts | 0 | 0 | 0 | 3
  Most Severe Ideation at Follow-up 4: Active Suicidal Ideation with Any Methods | 0 | 2 | 1 | 1
  Most Severe Ideation at Follow-up 4: Active Suicidal Ideation with Some Intent to Act | 1 | 1 | 1 | 0
  Most Severe Ideation at Follow-up 4: Active Suicidal Ideation with Specific Plan | 1 | 3 | 1 | 7
  Most Severe Ideation at Follow-up 5: number analyzed (Participants) | 34 | 37 | 24 | 31
  Most Severe Ideation at Follow-up 5: None | 25 | 23 | 12 | 15
  Most Severe Ideation at Follow-up 5: Wish to be Dead | 4 | 7 | 5 | 6
  Most Severe Ideation at Follow-up 5: Non-Specific Active Suicidal Thoughts | 1 | 2 | 0 | 2
  Most Severe Ideation at Follow-up 5: Active Suicidal Ideation with Any Methods | 2 | 1 | 5 | 4
  Most Severe Ideation at Follow-up 5: Active Suicidal Ideation with Some Intent to Act | 0 | 1 | 0 | 1
  Most Severe Ideation at Follow-up 5: Active Suicidal Ideation with Specific Plan | 2 | 3 | 2 | 3
  Most Severe Ideation at Follow-up 6: number analyzed (Participants) | 29 | 33 | 23 | 28
  Most Severe Ideation at Follow-up 6: None | 24 | 18 | 13 | 15
  Most Severe Ideation at Follow-up 6: Wish to be Dead | 2 | 8 | 3 | 5
  Most Severe Ideation at Follow-up 6: Non-Specific Active Suicidal Thoughts | 0 | 1 | 1 | 3
  Most Severe Ideation at Follow-up 6: Active Suicidal Ideation with Any Methods | 1 | 3 | 3 | 4
  Most Severe Ideation at Follow-up 6: Active Suicidal Ideation with Some Intent to Act | 0 | 1 | 0 | 0
  Most Severe Ideation at Follow-up 6: Active Suicidal Ideation with Specific Plan | 2 | 2 | 3 | 1

4. Primary Outcome: Columbia Suicide Severity Rating Scale Suicidal Ideation Intensity Scale Total Score
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) intensity subscale is the sum of 5 questions (frequency, duration, controllability, deterrents, and reasons for ideation) rated from 1-5, with 5 representing more severe intensity. Zero is entered if no suicidal ideation is reported. Total scores range from 0 to 25 with higher scores indicating more intense suicidal ideation.
Time Frame: Assessed at completion of inpatient treatment (average of 12 days), and on a monthly basis for 6 months follow-up.
Population: Data were missing due to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Presence of SUD With BCBT | Presence of SUD With TAU | Absence of SUD With BCBT | Absence of SUD With TAU
Number analyzed (Participants) | 52 | 56 | 38 | 41
score on a scale
  Intensity of Suicidal Ideation at Post-treatment | 6.04 (7.60) | 9.68 (7.94) | 6.84 (7.69) | 10.29 (8.32)
  Intensity of Suicidal Ideation at Follow-up 1: number analyzed (Participants) | 46 | 48 | 34 | 36
  Intensity of Suicidal Ideation at Follow-up 1 | 4.76 (7.55) | 7.79 (7.97) | 7.24 (7.11) | 9.42 (7.07)
  Intensity of Suicidal Ideation at Follow-up 2: number analyzed (Participants) | 42 | 47 | 30 | 35
  Intensity of Suicidal Ideation at Follow-up 2 | 4.48 (6.84) | 6.60 (7.45) | 8.23 (8.71) | 7.86 (8.67)
  Intensity of Suicidal Ideation at Follow-up 3: number analyzed (Participants) | 38 | 45 | 29 | 32
  Intensity of Suicidal Ideation at Follow-up 3 | 4.47 (6.78) | 6.76 (8.17) | 6.59 (7.78) | 6.81 (8.17)
  Intensity of Suicidal Ideation at Follow-up 4: number analyzed (Participants) | 37 | 39 | 27 | 34
  Intensity of Suicidal Ideation at Follow-up 4 | 2.35 (5.69) | 6.41 (7.30) | 7.19 (8.33) | 8.74 (8.37)
  Intensity of Suicidal Ideation at Follow-up 5: number analyzed (Participants) | 34 | 37 | 24 | 31
  Intensity of Suicidal Ideation at Follow-up 5 | 3.88 (6.68) | 5.68 (7.72) | 7.54 (8.28) | 7.87 (7.95)
  Intensity of Suicide Ideation at Follow-up 6: number analyzed (Participants) | 29 | 33 | 23 | 28
  Intensity of Suicide Ideation at Follow-up 6 | 2.83 (6.40) | 6.12 (7.29) | 6.91 (8.48) | 6.21 (7.15)

5. Primary Outcome: Number of Participants With Readmissions
Description: Readmission is determined using the participant's electronic medical record along with a self-report measure.
Time Frame: Assessed on a monthly basis for 6 months follow-up.
Population: Missing data are due to participants dropping out of the study during the follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Presence of SUD With BCBT | Presence of SUD With TAU | Absence of SUD With BCBT | Absence of SUD With TAU
Number analyzed (Participants) | 55 | 61 | 38 | 42
Participants
  Readmission at Follow-up 1 | 5 | 8 | 2 | 3
  Readmission at Follow-up 2 | 7 | 5 | 1 | 2
  Readmission at Follow-up 3 | 3 | 4 | 1 | 4
  Readmission at Follow-up 4: number analyzed (Participants) | 54 | 61 | 38 | 42
  Readmission at Follow-up 4 | 5 | 6 | 0 | 4
  Readmission at Follow-up 5: number analyzed (Participants) | 54 | 61 | 38 | 42
  Readmission at Follow-up 5 | 6 | 4 | 0 | 3
  Readmission at Follow-up 6: number analyzed (Participants) | 54 | 61 | 38 | 40
  Readmission at Follow-up 6 | 1 | 6 | 3 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the moment participants provided informed consent to the end of the 6-month follow-up period (approximately 7 months, dependent on length of inpatient stay).
Arm/Group | Presence of SUD With BCBT | Presence of SUD With TAU | Absence of SUD With BCBT | Absence of SUD With TAU
All-Cause Mortality (participants affected / at risk) | 1/62 | 1/65 | 0/41 | 0/45
Serious Adverse Events (participants affected / at risk) | 23/62 | 26/65 | 8/41 | 16/45
Other Adverse Events (participants affected / at risk) | 47/62 | 50/65 | 26/41 | 31/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Presence of SUD With BCBT (N=62) | Presence of SUD With TAU (N=65) | Absence of SUD With BCBT (N=41) | Absence of SUD With TAU (N=45)
Psychiatric Inpatient Hospitalization (Psychiatric disorders) | 12 (23) | 12 (19) | 6 (6) | 14 (17)
Change in Mental Health (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Change in Physical Health/Physical Injury (General disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 8 (12) | 10 (15) | 1 (2) | 4 (4)
Emergency Department Visit (General disorders) | 8 (10) | 4 (6) | 2 (2) | 2 (2)
Medical Hospitalization (General disorders) | 4 (4) | 5 (6) | 1 (1) | 2 (4)
Homelessness (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Presence of SUD With BCBT (N=62) | Presence of SUD With TAU (N=65) | Absence of SUD With BCBT (N=41) | Absence of SUD With TAU (N=45)
Change in Physical Health/Physical Injury (General disorders) | 26 (41) | 23 (34) | 20 (32) | 17 (23)
Reliable Change in Depression, Stress or Anxiety (Psychiatric disorders) | 8 (16) | 6 (7) | 6 (8) | 7 (15)
Change in Mental Health (Psychiatric disorders) | 22 (34) | 30 (47) | 18 (32) | 15 (32)
Suicide Attempt (Psychiatric disorders) | 7 (7) | 7 (7) | 2 (2) | 4 (6)
Emergency Department Visit (General disorders) | 30 (95) | 24 (66) | 8 (12) | 11 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT04168645/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04168645/ICF_001.pdf